CLINICAL TRIAL: NCT05543863
Title: Impact of Radial Distal Gastrectomy for Gastric Cancer on the Pharmacokinetics of Oral Antiplatelet Agents
Brief Title: Pharmacokinetics of Oral Antiplatelet Agents After Distal Gastrectomy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Kyungpook National University Chilgok Hospital (Other)
Responsible Party: Principal Investigator, Ji Yeon Park, Principle Investigator (Associate professor), Kyungpook National University Chilgok Hospital
Other Study IDs: KNUCH 2022-general-08
Record Dates: First submitted 2022-09-13; First posted 2022-09-16 (Actual); Last update posted 2022-09-21 (Actual); Status verified 2022-09

CONDITIONS: Stomach Neoplasm; Cardiovascular Diseases; Cerebrovascular Disease
MeSH Terms: conditions — Stomach Neoplasms; Cardiovascular Diseases; Cerebrovascular Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Biospecimen Retention: Samples With DNA — blood samples
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Platelet function testing — platelet function testing (Platelet function analyzer-100 (PFA-100) collagen epinephrine closure time, VerifyNowⓇ Assays (aspirin, P2Y12)) before surgery and 5 days, 3 months after surgery

SUMMARY:
This study is aimed to investigate the changes in pharmacokinetics and efficacy of antiplatelet agents before and after distal gastrectomy in gastric cancer patients taking oral antiplatelet agents for primary or secondary treatment for cardiovascular disease and to evaluate its impact on the occurrence of postoperative bleeding complications and thromboembolic events.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with pathologically proven gastric cancer of clinical stage I according to the AJCC 8th edition.
* Patients who are scheduled to undergo distal gastrectomy (access: either minimally invasive surgery or open surgery)
* Patients taking aspirin and/or clopidogrel for primary or secondary prevention for cardiovascular disease or cerebrovascular disease before surgery.
* age 18 - 90 years
* A person who voluntarily agrees to participate in this study and signs the consent form.

Exclusion Criteria:

* Patients with coagulation disorder or abnormal findings in coagulation test (low platelet count, prolonged PT/aPTT)
* Patients taking other anticoagulants in combination
* Patients with imparied liver or renal function that may affect drug metabolism.

Impaired liver function: liver cirrhosis Impaired renal function: CKD grade 3 or higher

* Patients requiring adjuvant chemotherapy after surgery that may affect postoperative bone marrow function and hematopoietic function (those with gastric cancer of clinical stage II or more according to the AJCC 8th edition)
* Patients participating in other clinical trials within 6 months
* Vulnerable patients (pregnant women, those with cognitive impairment, etc)

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are taking antiplatelet agents and scheduled for distal gastrectomy for gastric cancer
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2022-08-20 (Actual); Primary Completion 2023-03-31 (Estimated); Study Completion 2023-05-31 (Estimated)

PRIMARY OUTCOMES:
platelet function testing at 5 days | 5 days
  Difference in the platelet function testing results between before and 5 days after surgery.

SECONDARY OUTCOMES:
Platelet function testing at 3 months | 3 months
  Difference in the platelet function testing results between before and 3 months after surgery
postoperative complications | 3 months
  ■ incidence of postoperative bleeding and thromboembolic events within 3 months after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Ji Yeon Park, MD, Principal Investigator — Dept. of Surgery, Kyungpook National Univ. Chilgok Hosptal
Locations (1):
- Dept. of Surgery, Kyungpook National University Chilgok Hospital, Daegu, South Korea

IPD SHARING:
Plan to Share IPD: No